CLINICAL TRIAL: NCT02492061
Title: Demand Creation for Couples' HIV Counseling and Testing, Linkage to and Retention in HIV Care Among Married Couples in Rakai, Uganda
Brief Title: Demand Creation for Couples' HIV Counseling and Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Rakai Health Sciences Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/HD07/18256U
Record Dates: First submitted 2015-06-14; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: HIV/AIDS
Keywords: couples' HCT married couples; Rakai; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Demand creation (Active Comparator): In the intervention arm, demand creation for couples' HCT is done using small group (comprising about 20 people), couple-focused or men-only, interactive sessions. A senior counselor facilitates the sessions in which the advantages and fears associated with couples' HCT are discussed with invited couples or men. The sessions are reinforced by testimonies from couples or men who have ever tested as a couple. Attending couples or men receive couple invitation coupons inviting them to test for HIV together with their partners at a designated health facility in the community.
  Interventions: Behavioral: Demand creation for couples' HCT
- Standard of care (No Intervention): In the standard of care arm, participants receive general adult health talks to educate them about the importance of HIV testing (including couples' HCT) but no invitations are issued to invite couples to test for HIV together with their partners at a designated health facility. However, couples can seek HCT out of their own volition. The sessions are not stratified by marital status, and attendants include all those who are willing and are able to attend.

INTERVENTIONS:
Behavioral: Demand creation for couples' HCT — The demand creation for couples' HCT intervention aims at improving uptake of couples' HCT among married couples in Rakai, southwestern Uganda
  Arms: Demand creation

SUMMARY:
This study aims at assessing the effect of a demand-creation intervention on couples' HIV counseling and testing (couples' HCT) uptake among married couples who have never tested together as a couple. The study is being implemented in 12 clusters; six intervention and six comparison clusters. A total of 1,538 couples will be enrolled into the study; 769 couples per arm. Couples in the intervention communities are invited to participate in small group, couple-focused or men-only, interactive sessions lasting 3-4 hours in which the advantages and fears associated with couples' HCT are discussed with invited couples to motivate them to consider testing together as a couple. The meetings are reinforced with testimonies from previously tested couples. At the end of the sessions, couples or men receive invitation coupons which they present to a designated health facility to receive couples' HCT services (couples are free to receive individual HCT or not to honor the invitation, if they are not interested in taking the HCT offer). In the comparison communities, standard of care health education activities including general adult community sessions are held but couples do not receive any invitations to test as a couple. Nevertheless, couples in the comparison communities have unlimited access to HIV counseling and testing services that are offered by the Rakai Health Sciences Program within the study communities. The investigators hypothesize that couples in the intervention arm will be more likely to test together than those in the comparison arm. The study objectives include: a) exploring the motivations for and barriers to couples' HCT uptake; b) assessing the effect of a demand-creation intervention on couples' HCT uptake among married couples with no prior couples' HCT experience, and c) exploring the effect of couples' HCT vs. individual HCT on linkage to and retention in HIV care.

DETAILED DESCRIPTION:
This is a cluster-randomized intervention trial aimed at assessing the effect of a community-based demand creation intervention on couples' HIV counseling and testing (couples' HCT) among 1,538 married couples with no prior couples' HCT experience, resident in three study regions/clusters in Rakai district. The study population is composed of couples in which both partners have never received couples' HCT. The intervention utilizes couple-focused meetings and men-only meetings to promote couples' HCT while invitation coupons are issued to all targeted couples inviting them to come for couples' HCT at designated health facilities within Rakai district. Initially, a qualitative sub-study was implemented to explore the motivations for and barriers to couples' HCT uptake - these aspects are important for the design of the intervention. This was followed by a baseline study to document the current levels of HCT uptake in the community, and then the intervention implementation followed suit. The study was implemented in 12 study communities; 6 of which served as the intervention while the other 6 served as comparison communities. Data collection for the post-intervention survey was completed in April 2015. Efforts are currently underway to assess linkage to and retention in HIV care among couples that tested as a result of the campaign.

The study has 3 inter-related sub-studies (objectives), namely: (i) Exploring the motivation for and barriers to couples' HCT uptake at community level (b) Assessing the effect of a demand creation intervention on couples' HCT uptake among married couples with no prior couples' HCT, and (c) Determining the effect of couples' HCT relative to individual HCT on linkage to and retention in HIV care among HIV-positive and HIV-discordant couples that are not yet in HIV care. Sub-study I comprises use of qualitative research methods to explore the motivation for and barriers to couples' HCT uptake through 18 focus group discussions (FGDs) and 12 key informant interviews. Findings from this sub-study helped to inform the design of a demand-creation HCT intervention aimed at improving couples' HCT uptake in selected communities in Rakai. Sub-study II is a one-year community intervention trial aimed at assessing the effect of a demand-creation intervention (comprising couple-focused meetings; couple invitation coupons; and men-only sensitization meetings) on couples' HCT uptake among couples with no prior couples' HCT experience. The study will be implemented in 3 study regions with differing HIV prevalence levels (low (9.7-11.2%), middle (11.4-16.4%) and high (20.5-43%)) in Rakai district. Overall, 1,538 eligible couples were invited to participate in the baseline study. Of these, 2,135 were interviewed at baseline and followed up 12 months later. In sub-study III, the investigators will enroll 462 couples in which at least one partner is HIV-positive and follow them up for 1, 3 and 6 months after HIV diagnosis to determine the effect of couples' HCT [vis-à-vis individual HCT] on timely linkage to and retention in HIV care.

To estimate the sample size for the intervention, the investigators assumed a minimum improvement in couples' HCT uptake of 10% in the intervention communities compared with a baseline of 25% in the standard of care/comparison communities (Grabowski et al. 2014). The investigators set two-sided alpha level at 0.05 and assumed a power of 90% to detect differences in the proportion of couples accepting couples' HCT between the intervention and comparison communities. The investigators used 12 study communities/clusters and accounted for cluster design effect using an intra-class correlation of 0.0039 based on an earlier study in Rakai (Todd et al. 2003). Based on these assumptions, the investigators estimated that they would need to enroll 769 couples in each arm (i.e. intervention and comparison communities), after adjusting for non-response rate (out-migration, refusal to participate, and loss to follow-up) estimated at 15% (Gray et al. 2007). The final sample was 1,538 couples (or 3,076 individuals). Sample size estimation was done using the sampsi and sampclus commands in STATA (STATA statistical software, version 11.2).

ELIGIBILITY:
Inclusion Criteria:

* Currently married individuals
* Marital duration of >=1 year
* No previous HIV testing or previous individual HIV testing
* If HIV-positive, not yet enrolled in HIV care

Exclusion Criteria:

* Not currently married
* Marital duration < 1 year
* Previous receipt of couples' HIV counseling and testing
* Previous self-reported joint HIV status disclosure

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3076 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of married individuals who have received couples' HCT | 3 months after end of intervention
  Overall proportion of married individuals that will have received couples' HCT (out of those who have never received couples' HCT) as a result of the intervention. We will compare the proportion of married individuals receiving couples' HCT in the intervention arm to the proportion receiving couples' HCT in the comparison arm. The intervention will be considered to have been successful if the proportion of married individuals who received couples' HCT is 10% higher in the intervention than in the comparison arm.

SECONDARY OUTCOMES:
Proportion of HIV-positive individuals who have been enrolled in HIV care | 6 months after end of intervention
  Proportion of HIV-positive individuals (who were not yet in HIV care) who have been enrolled in HIV care at 1, 3 and 6 months after the intervention. We will assess differences in enrollment in HIV care between those who received couples' HCT and those who received individual HCT to determine the relative effect of couples' HCT over individual HCT in improving linkage to HIV care.
Proportion of enrolled HIV-positive individuals who have been retained in HIV care | 9 months after end of intervention
  Proportion of enrolled HIV-positive individuals who are still in HIV care at 3, 6, and 9 months after enrollment. We will assess differences in retention in HIV care between those who previously received couples' HCT (prior to enrollment) and those who previously received individual HCT to determine the relative effect of couples' HCT over individual HCT in improving retention in HIV care.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph KB Matovu, MHS, Principal Investigator — Makerere University

REFERENCES:
- [Background] Grabowski MK, Lessler J, Redd AD, Kagaayi J, Laeyendecker O, Ndyanabo A, Nelson MI, Cummings DA, Bwanika JB, Mueller AC, Reynolds SJ, Munshaw S, Ray SC, Lutalo T, Manucci J, Tobian AA, Chang LW, Beyrer C, Jennings JM, Nalugoda F, Serwadda D, Wawer MJ, Quinn TC, Gray RH; Rakai Health Sciences Program. The role of viral introductions in sustaining community-based HIV epidemics in rural Uganda: evidence from spatial clustering, phylogenetics, and egocentric transmission models. PLoS Med. 2014 Mar 4;11(3):e1001610. doi: 10.1371/journal.pmed.1001610. eCollection 2014 Mar. PMID 24595023
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Todd J, Carpenter L, Li X, Nakiyingi J, Gray R, Hayes R. The effects of alternative study designs on the power of community randomized trials: evidence from three studies of human immunodeficiency virus prevention in East Africa. Int J Epidemiol. 2003 Oct;32(5):755-62. doi: 10.1093/ije/dyg150. PMID 14559745
- [Derived] Matovu JK, Todd J, Wanyenze RK, Kairania R, Serwadda D, Wabwire-Mangen F. Evaluation of a demand-creation intervention for couples' HIV testing services among married or cohabiting individuals in Rakai, Uganda: a cluster-randomized intervention trial. BMC Infect Dis. 2016 Aug 8;16:379. doi: 10.1186/s12879-016-1720-y. PMID 27502776